CLINICAL TRIAL: NCT04184752
Title: Urodynamically Age-specific Prevalence of Detrusor Underactivity and Bladder Outlet Obstruction in Female Voiding Dysfunction Without Cystocele
Brief Title: Prevalence of Detrusor Underactivity and Bladder Outlet Obstruction in Female Without Cystocele
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201907011RINC
Record Dates: First submitted 2019-11-28; First posted 2019-12-04 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2019-08

CONDITIONS: Voiding Disorders
Keywords: Bladder outlet obstruction; Detrusor underactivity; Voiding dysfunction
MeSH Terms: conditions — Urinary Bladder Neck Obstruction; Urinary Bladder, Underactive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Detrusor underactivity: The DU was defined when the PdetQmax was less than 20 cmH2O, the Qmax was less than 15 mL/s, and the bladder voiding efficiency (BVE) was less than 90 %. BVE = voided volume / (voided volume+ PVR) x 100%.
  Interventions: Diagnostic Test: Urodynamic study
- Bladder outlet obstruction: The BOO was defined when the PdetQmax was not less than 40 cmH2O, and the Qmax was less than 12 mL/s.
  Interventions: Diagnostic Test: Urodynamic study
- Non-DU/BOO group: Those women without DU or BOO were allocated to the non-DU/BOO group.
  Interventions: Diagnostic Test: Urodynamic study

INTERVENTIONS:
Diagnostic Test: Urodynamic study — The urodynamic assessment included uroflowmetry, filling cystometry with 35°C distilled water at a rate of 60 mL/sec, a pressure flow study, and a stress urethral pressure profile with patient in sitting position [14]. A 20-minute pad test for each woman was also performed [15, 16]. Multichannel urodynamic equipment (Life-Tech, Houston, TX, USA) with computer analysis and Urovision (Urolab Janus System V, Houston) was used. All terminology conformed to the standards recommended by the ICS [3]. All procedures were performed by an experienced technician, and the data were interpreted by a single observer to avoid interobserver variability.
  Other Names: Pad test

SUMMARY:
Women with symptoms of voiding dysfunction may be associated with detrusor underactivity (DU) or bladder outlet obstruction (BOO). The treatment strategies are different between DU and BOO. In general, urodynamic/videourodynamic studies are important for differential diagnosis. However, urodynamic/videourodynamic studies are invasive. The investigators are interested in whether there were specific symptoms or measurements that can be used for initial differential diagnosis between DU and BOO. Thus, the aim of this study was to elucidate the prevalence of DU and BOO in each age group and elucidate the clinical and urodynamic differences between the DU, BOO and non-DU/BOO groups.

DETAILED DESCRIPTION:
Between April 1996 and September 2018, all women with symptoms of voiding dysfunction who visited the urogynecological department of a medical center for urodynamic evaluation were reviewed. Those women who have no complete data of maximum flow rate (Qmax), voided volume, post-void residual volume (PVR) and detrusor pressure at a maximum flow rate (PdetQmax) were excluded from this study. Besides, women with cystocele were also excluded. The DU was defined when the PdetQmax was less than 20 cmH2O, the Qmax was less than 15 mL/s, and the bladder voiding efficiency (BVE) was less than 90 %. The BOO was defined when the PdetQmax was not less than 40 cmH2O, and the Qmax was less than 12 mL/s. BVE = voided volume / (voided volume+ PVR) x 100%. Those women without DU or BOO were allocated to the non-DU/BOO group.

STATA software was used for statistical analysis. ANOVA test with Bonferroni correction or chi-square test was used for statistical analysis as appropriate. Linear regression analysis with age adjustment was used to assess the adjusted effect of variables. P < 0.05 was considered as statistical significant.

ELIGIBILITY:
Inclusion Criteria:

* Women with symptoms of voiding dysfunction.

Exclusion Criteria:

* Cystocele
* Those women who have no complete data of maximum flow rate (Qmax), voided volume, post void residual volume (PVR) and detrusor pressure at maximum flow rate (PdetQmax) were excluded from this study.

Ages: 20 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All women with symptoms of voiding dysfunction and without cystocele who visited the urogynecological department of a medical center for urodynamic evaluation were reviewed.
Sampling Method: Non-Probability Sample
Enrollment: 602 (Actual)
Dates: Start 1996-04-01 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Detrusor underactivity or Bladder outlet obstruction | Between April 1996 and September 2018
  The DU was defined when the PdetQmax was less than 20 cmH2O, the Qmax was less than 15 mL/s, and the bladder voiding efficiency (BVE) was less than 90 %. The BOO was defined when the PdetQmax was not less than 40 cmH2O, and the Qmax was less than 12 mL/s. BVE = voided volume / (voided volume+ PVR) x 100%.

CONTACTS AND LOCATIONS:
Overall Officials: Ho-Hsiung Lin, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available to other researchers.

REFERENCES:
- [Result] Haylen BT, de Ridder D, Freeman RM, Swift SE, Berghmans B, Lee J, Monga A, Petri E, Rizk DE, Sand PK, Schaer GN. An International Urogynecological Association (IUGA)/International Continence Society (ICS) joint report on the terminology for female pelvic floor dysfunction. Int Urogynecol J. 2010 Jan;21(1):5-26. doi: 10.1007/s00192-009-0976-9. Epub 2009 Nov 25. PMID 19937315
- [Result] Choi YS, Kim JC, Lee KS, Seo JT, Kim HJ, Yoo TK, Lee JB, Choo MS, Lee JG, Lee JY. Analysis of female voiding dysfunction: a prospective, multi-center study. Int Urol Nephrol. 2013 Aug;45(4):989-94. doi: 10.1007/s11255-013-0475-2. Epub 2013 May 31. PMID 23722818
- [Result] Karmakar D, Sharma JB. Current concepts in voiding dysfunction and dysfunctional voiding: A review from a urogynaecologist's perspective. J Midlife Health. 2014 Jul;5(3):104-10. doi: 10.4103/0976-7800.141185. PMID 25316994 (Retraction: PMID 29628732 J Midlife Health. 2018 Jan-Mar;9(1):50)
- [Result] Robinson D, Staskin D, Laterza RM, Koelbl H. Defining female voiding dysfunction: ICI-RS 2011. Neurourol Urodyn. 2012 Mar;31(3):313-6. doi: 10.1002/nau.22213. Epub 2012 Mar 13. PMID 22415792
- [Result] Hsiao SM, Lin HH, Kuo HC. Videourodynamic Studies of Women with Voiding Dysfunction. Sci Rep. 2017 Jul 28;7(1):6845. doi: 10.1038/s41598-017-07163-2. PMID 28754926
- [Result] Lukacz ES, DuHamel E, Menefee SA, Luber KM. Elevated postvoid residual in women with pelvic floor disorders: prevalence and associated risk factors. Int Urogynecol J Pelvic Floor Dysfunct. 2007 Apr;18(4):397-400. doi: 10.1007/s00192-006-0164-0. Epub 2006 Jun 28. PMID 16804634
- [Result] Milleman M, Langenstroer P, Guralnick ML. Post-void residual urine volume in women with overactive bladder symptoms. J Urol. 2004 Nov;172(5 Pt 1):1911-4. doi: 10.1097/01.ju.0000140502.34334.75. PMID 15540753